CLINICAL TRIAL: NCT04260217
Title: A Phase Ib /II Open-label, Multi-center Study to Evaluate the Safety, Tolerability and Efficacy of APG-2575 Single Agent or in Combination With Ibrutinib or Rituximab in Patients With Waldenström Macroglobulinemia (MAPLE-1)
Brief Title: APG-2575 Single Agent or in Combination With Ibrutinib or Rituximab in Patients With Waldenström Macroglobulinemia
Acronym: MAPLE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575WU101
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Lisaftoclax

STUDY DESIGN:
Intervention Model Description: APG2575 400 mg ramp up arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APG2575 400 mg (Experimental): APG2575 400mg ramp up arm
  Interventions: Drug: APG2575 400 mg; Drug: APG2575 600 mg; Drug: APG2575 800 mg
- APG2575 600 mg (Experimental): APG2575 600 mg ramp up arm
  Interventions: Drug: APG2575 600 mg; Drug: APG2575 800 mg
- APG2575 800 mg arm (Experimental): APG2575 800 mg arm ramp up
  Interventions: Drug: APG2575 800 mg

INTERVENTIONS:
Drug: APG2575 400 mg — APG2575 400 mg
  Arms: APG2575 400 mg
Drug: APG2575 600 mg — APG2575 600 mg
  Arms: APG2575 400 mg; APG2575 600 mg
Drug: APG2575 800 mg — APG2575 800 mg

SUMMARY:
Phase Ib/II study of safety, tolerability, efficacy and PK of APG-2575 as a single agent or in combination with other therapeutic agents including ibrutinib or rituximab.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase Ib/II study of safety, tolerability, efficacy and PK of APG-2575 as a single agent or in combination with other therapeutic agents including ibrutinib or rituximab. The study consists of the dose escalation and the dose expansion phases. The clinical trial will have multiple arms with ability to subsequently add more treatment arms based upon clinical activity of APG2575 in WM. Initially the study will contain 3 arms noted below, all the arms are independent.

Arm A: APG-2575 will be administered as a single agent to determine the MTD/RP2D in subjects who are relapsed/resistant or intolerant to ibrutinib or other BTK inhibitors.

The Dose escalation phase of APG-2575 as monotherapy will use mTPI-2 design. The starting target dose (using ramp-up if needed) is 400 mg (dose level; DL1) and will be increased to 600 mg (DL2), 800 mg (DL3) accordingly. Doses can be increased to higher level depending on safety and PK results based on discussions of the Investigators and Sponsor. APG-2575 will be administered orally once daily until time of progression or unacceptable toxicity. After the MTD/RP2D is determined, up to 12 additional patients will be enrolled at RP2D in dose-expansion phase to further evaluate safety and efficacy of APG-2575.

Arm B: APG-2575 will be administered in combination with ibrutinib in subjects with previously untreated WM.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Local confirmed clinicopathological diagnosis of WM in accordance with the consensus panel of the Second International Workshop on WM (Owen 2003).
2. WM patients with symptomatic and measurable disease (defined as presence of serum immunoglobulin M (IgM)>0.5g/dL), requiring treatment as per mSMART guidelines (Kyle 2003): with B symptoms (fever, night sweats, fatigue, night sweats weight loss), progressive lymphadenopathy or splenomegaly, anemia (hemoglobin value of <10 g/dL) or platelet count <100*109/L due to marrow infiltration. Complications such as hyperviscosity syndrome, symptomatic sensorimotor peripheral neuropathy due to WM, systemic amyloidosis related to WM, renal insufficiency related to WM, or symptomatic cryoglobulinemia may also be indications for therapy.
3. For Arm A only: Have received at least one prior therapy for WM. Patient must have either failed (defined as progressing while on or within 6 months of treatment with ibrutinib treatment) or intolerant to ibrutinib.
4. For Arm B only: Previously untreated WM.
5. For Arm C only: Have received at least one prior therapy, relapsed or refractory WM.
6. Adequate hematologic function defined as:

   1. ANC ≥1.0 x 109/L independent of growth factor support within 7 days of the first dose with study drug.
   2. Hemoglobin ≥9 g/dL without transfusion or growth factor support within 7 days of the first dose of study drug.
   3. Platelet count ≥ 75 x 109/L without transfusion support within 7 days of the first dose of study drug.
7. Adequate hepatic and renal function defined as:

   1. AST and ALT < 2.5 x ULN (upper limit of normal)
   2. Glomerular filtration rate (GFR) >30mL/min
   3. Bilirubin< 1.5 x ULN
8. PT/INR ≤1.5 x ULN and PTT (aPTT) ≤1.5 x ULN.
9. ≥18 years of age.
10. Eastern Cooperative Oncology Group (ECOG) ≤1.
11. Life expectancy≥3 months.
12. Female subjects who are of non-reproductive potential (i.e., post-menopausal by history-no menses for ≥2 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
13. Male and female subjects who agree to use highly effective methods of birth control (e.g.,condoms, implants, injectables, combined oral contraceptives, some intrauterine devices[IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for 30 days after the last dose of study drug and 90 days (males) after the last dose of study drug.

Symptomatic disease meeting at least 1 of the recommendations from the Second International Workshop on Waldenström Macroglobulinemia for requiring treatment (Kyle 2003):

1. Constitutional symptoms documented in the subject's chart with supportive objective measures, as appropriate, defined as one or more of the following disease-related symptoms or signs:

   1. Unintentional weight loss ≥10% within the previous 6 months prior to Screening
   2. Fevers higher than 100.5°F or 38.0°C for 2 or more weeks prior to Screening without evidence of infection
   3. Night sweats for more than 1 month prior to Screening without evidence of infection
2. Clinically relevant fatigue which is not relieved by rest due to WM
3. Symptomatic hyperviscosity or serum viscosity levels greater than 4.0 centipoises
4. Lymphadenopathy which is either symptomatic or bulky (≥5cm in maximum diameter)
5. Symptomatic hepatomegaly and/or splenomegaly and/or organ tissue infiltration
6. Peripheral neuropathy due to WM
7. Symptomatic cryoglobulinemia
8. Cold agglutinin anemia
9. IgM related immune hemolytic anemia and/or thrombocytopenia
10. Nephropathy related to WM
11. Amyloidosis related to WM
12. Hemoglobin ≤10g/dL
13. Platelet count <100 x109/L
14. Serum monoclonal protein >5g/dL, with or without overt clinical symptoms.
15. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Exclusion Criteria:

* Criteria for exclusion:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. For Arm A only: Patients who have never been treated with ibrutinib.
2. For Arm B only: Patients who have previously received any treatment for WM.
3. For Arm C only:

   1. Patients who have previously been treated with ibrutinib or other BTK inhibitor.
   2. Disease that is refractory to the last prior rituximab based-therapy defined as either Relapse after the last rituximab-based therapy (<12 months since last dose of rituximab), OR Failure to achieve at least a MR after the last rituximab-based therapy.
   3. Rituximab treatment within the last 12 months before the first dose of study drug.
   4. Known anaphylaxis or IgE-mediated hypersensitivity to murine proteins or to any component of rituximab.
4. Patients with central nervous system involvement (Bing-Neel syndrome), active infection (including active hepatitis B or C virus infection, known human immunodeficiency virus (HIV) positive) or any other serious (unresolved) medical condition.
5. Plasmapheresis <35 days prior to the initiation of study drug. (Note: Subjects with high IgM values or hyper-viscosity symptoms during screening may receive plasmapheresis prior to initiating study drug if the previous plasmapheresis was performed >35 days before the plasmapheresis performed during screening (in order to obtain a true baseline IgM value for efficacy evaluations).
6. Failure to have fully recovered (i.e., ≤Grade 1 toxicity) from the reversible effects of prior treatment for WM.
7. Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) ≥470 msec.
8. Unable to swallow tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
9. History of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) defined by positive polymerase chain reaction (PCR).
10. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
11. Major surgical procedure within ≤14 days prior to initiating study treatment, or anticipation of the need for major surgery during the course of the study treatment, radiotherapy ≤14 days prior to initiating study treatment, systemic treatment within 14 days before the first dose of APG-2575.
12. Recent infection requiring systemic treatment that was completed≤14 days before the first dose of study drug.
13. Any uncontrolled active systemic infection.
14. Any concurrent malignancy.
15. Concomitant use of warfarin or other Vitamin K antagonists (eg. phenoprocoumon).
16. Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor.
17. Known bleeding disorders (eg, von Willebrand's disease) or hemophilia.
18. History of stroke or intracranial hemorrhage within 12 months prior to enrollment.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Primary Toxicity Endpoint: dose limiting toxicity (DLT) | 42 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 6 weeks (2 cycles) of study treatment. These will be assessed via CTCAE version 5.0
Maximally tolerated dose (MTD) | 42 days
  MTD will be determined based on DLTs observed during the first 6 weeks (2 cycles) of study treatment

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Weill Cornell Univ Hospitals, New York, New York
  - MD Anderson, Houston, Texas
- St. Vincent Hospital, Melbourne, Australia
- China (8):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Chaoyang Hospital, Beijing
  - The First Affiliated Hospital,College Of Medicine,Zhejiang University, Hangzhou
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - The First Affiliated Hospital Of Soochow University, Suzhou
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin
  - Henan Cancer Hospital, Zhengzhou